CLINICAL TRIAL: NCT00001029
Title: A Randomized, Double-Blind, Three-Arm Study Comparing Combination to Monthly Alternating Nucleoside Therapy for the Treatment of Advanced HIV Disease (CD4 <= 50/mm3) With a Prior History of Nucleoside Therapy
Brief Title: A Comparison of Three Treatments for Advanced HIV Disease in Patients Who Have Received Nucleoside Therapy in the Past
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 193; 11168 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; Zalcitabine; Didanosine

INTERVENTIONS:
Drug: Zidovudine
Drug: Zalcitabine
Drug: Didanosine

SUMMARY:
To compare the efficacy, safety and tolerance, and other clinical and immunologic effects of zidovudine (AZT) plus zalcitabine (dideoxycytidine; ddC), AZT plus didanosine (ddI), and AZT alternating monthly with ddI as measured by differences in survival among HIV-infected persons who have received 6 or more months of nucleoside monotherapy and have a CD4 count greater than or equal to 50 cells/mm3.

Combining two nucleoside drugs has the theoretical advantage of optimal protection against the evolution of resistant strains of HIV. However, one major problem with combination nucleoside therapy in patients with advanced disease is the increased toxicity resulting from such therapy. One approach to minimize toxicity while perhaps retaining some of the benefits of combination therapy is to alternate the two drugs.

DETAILED DESCRIPTION:
Combining two nucleoside drugs has the theoretical advantage of optimal protection against the evolution of resistant strains of HIV. However, one major problem with combination nucleoside therapy in patients with advanced disease is the increased toxicity resulting from such therapy. One approach to minimize toxicity while perhaps retaining some of the benefits of combination therapy is to alternate the two drugs.

Patients are randomized to one of three treatment arms: AZT plus ddI, AZT plus ddC, and AZT alone alternating monthly with ddI. Half of the patients receiving AZT alternating monthly with ddI will start with AZT, while the other half will start with ddI. Treatment continues until death or termination of the study. Patients are followed every 4 weeks. The study will include a subset of patients for whom virologic, pharmacokinetic, and macroneurologic assessments will be made.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* PCP prophylaxis.

Allowed:

* Erythropoietin.
* Prophylaxis for MAI or fungal infections.
* Antibiotics.
* Over-the-counter, alternative, or regularly prescribed drugs.
* Steroids, if for < 21 days.

Concurrent Treatment:

Allowed:

* Radiation therapy for cutaneous Kaposi's sarcoma.

Patients must have:

* HIV infection.
* CD4 count <= 50 cells/mm3.
* Prior nucleoside monotherapy for at least 6 months.
* Life expectancy of at least 6 months.

Prior Medication: Required:

* Nucleoside monotherapy for at least 6 months. Active alcohol or drug abuse.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Severe peripheral neuropathy.
* Psychological or emotional problems sufficient to prevent study compliance.

Concurrent Medication:

Excluded:

* Systemic chemotherapy for malignancy.
* Acute or induction therapy for opportunistic infection.

Patients with the following prior conditions are excluded:

* History of acute or chronic pancreatitis.
* Grade 3 or greater toxicity to AZT, ddI, or ddC on two or more occasions.

Prior Medication:

Excluded:

* Non-study nucleosides or biologic response modifiers within 7 days prior to study entry.
* Acute therapy for opportunistic process within 14 days prior to study entry.
* Acute systemic therapy for other medical conditions within 14 days prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 654
Dates: Study Completion 1993-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: WK Henry, Study Chair; JO Kahn, Study Chair; HH Balfour, Study Chair
Locations (37):
- United States (35):
  - USC CRS, Los Angeles, California
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Northwestern University CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Hennepin County Med. Ctr., Div. of Infectious Diseases, Minneapolis, Minnesota
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell University A2201, New York, New York
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico
- Mbeya Med. Research Program, Mbeya Referral Hosp. CRS, Mbeya, Tanzania

REFERENCES:
- [Background] Fichtenbaum CJ, Powderly WG. Refractory mucosal candidiasis in patients with human immunodeficiency virus infection. Clin Infect Dis. 1998 Mar;26(3):556-65. doi: 10.1086/514571. PMID 9524822
- [Background] Henry K, Tierney C, Kahn J, Balfour H, Jiang Q, Kmack A, Fischl M. A randomized, double-blind, placebo-controlled study comparing combination nucleoside and triple therapy for the treatment of advanced HIV disease (CD4 less than or equal to 50/mm(3)). Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:207 (abstract no LB6)
- [Background] Henry K, Erice A, Tierney C, Balfour HH Jr, Fischl MA, Kmack A, Liou SH, Kenton A, Hirsch MS, Phair J, Martinez A, Kahn JO. A randomized, controlled, double-blind study comparing the survival benefit of four different reverse transcriptase inhibitor therapies (three-drug, two-drug, and alternating drug) for the treatment of advanced AIDS. AIDS Clinical Trial Group 193A Study Team. J Acquir Immune Defic Syndr Hum Retrovirol. 1998 Dec 1;19(4):339-49. doi: 10.1097/00042560-199812010-00004. PMID 9833742